CLINICAL TRIAL: NCT02333227
Title: Saving Lives at Birth: Primary Prevention of Periodontal Disease in Relation to Preterm Birth in Malawi (Prevention of Prematurity and Xylitol)
Brief Title: Saving Lives at Birth: Primary Prevention of Periodontal Disease in Relation to Preterm Birth in Malawi
Acronym: PPaX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kjersti Aagaard, Associate Professor and Vice Chair of Research, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHSRC # 1030; H-35933 (Other: Baylor College of Medicine)
Record Dates: First submitted 2014-12-23; First posted 2015-01-07 (Estimated); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Preterm Birth; Periodontal Disease; Caries, Dental
MeSH Terms: conditions — Premature Birth; Periodontal Diseases; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Cluster of sites not receiving xylitol gum. This is a cluster randomized trial, whereby 4 sites will not receive the intervention of xylitol gum in the prepregnancy and early pregnancy interval.
- Xylitol (Experimental): Cluster of sites receiving xylitol gum.
  Interventions: Dietary Supplement: Xylitol gum

INTERVENTIONS:
Dietary Supplement: Xylitol gum — This is a cluster randomized trial, whereby 4 sites will receive the intervention of xylitol gum in the prepregnancy and early pregnancy interval.
  Arms: Xylitol

SUMMARY:
The hypothesis of the investigators' project is that comprehensive primary preterm birth prevention, inclusive of maternal oral health with xylitol chewing gum (the intervention), will reduce the rate of periodontal disease and caries, preterm birth prevalence, and neonatal mortality.

DETAILED DESCRIPTION:
Significance and Impact: Adverse birth outcomes related to the length of gestation (preterm birth) are recognized as one of the most significant disorders in maternal-child health at a global scale. In the developed world, the preterm birth rate approximates 7%. In Malawi, the investigators have recently demonstrated that this rate more than triples to approximate 26.1%. Of the 4 million newborn deaths annually, nearly 1/3 (27%) are directly attributable to prematurity with another 36% secondary to related opportunistic infections (sepsis, pneumonia, gastrointestinal). 75% of the 4 million deaths occur within the first week of life, with the vast majority occurring in the first 48 hours. For those that do survive, there are persistent and lifelong risks due to stunted growth, chronic infection, retinopathy of prematurity, and bronchopulmonary dysplasia. The link between maternal oral health (periodontal disease in particular) and risk of preterm birth has been demonstrated across all populations (rural and urban, in both industrialized and developing regions) studied to date. However, in multiple randomized controlled trials treatment of active periodontal disease with scaling and planning during pregnancy has failed to demonstrate a significant benefit in preventing preterm birth.

Why would maternal oral health impact preterm birth? In rodents, subcutaneous inoculations with periodontal pathogens cause dose-dependent decreases in pup weights, and elicit inflammatory responses that can trigger preterm birth when present in amniotic fluid. Periodontitis (defined as a destructive inflammation of the periodontium) has a prevalence of 30% or greater in women of child bearing age. By definition, it involves microbial infiltration of the periodontium, which stimulates a chronic inflammatory response, recurrent bacteremia, and the production of cytokines and prostaglandins which trigger risk of preterm birth. It is the same production of prostaglandins which are felt to mediate the risk of preterm birth. So if the investigators know that there is biologic evidence that periodontitis is related to preterm birth, but treating active periodontitis does not reduce these morbidities, is it possible that preventing periodontitis might prevent preterm birth and low birth weight? If so, what are the least expensive efficacious preventative measures? The investigators' overarching hypothesis is that comprehensive primary preterm birth prevention, inclusive of maternal oral health with xylitol chewing gum (the intervention), will reduce the rate of periodontal disease and caries, preterm birth prevalence, and neonatal mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment at <20 weeks gestation by best obstetrical estimate, or
2. Enrollment post partum with an anticipated next pregnancy within 18 months, or
3. Enrollment preconception with an anticipated pregnancy within 18 months (preconception); and
4. Cognitively aware enough to participate in the study
5. >18 years of age (in Malawi, constitutes a legal adult and capacity to consent for study)
6. Willing to participate in the study
7. Willing to undergo at least two periodontal exams
8. Willing to chew 1 piece of xylitol gum for 10 minutes after the morning and evening meal (intervention sites)
9. Anticipating to remain within the region for 18 months

Exclusion Criteria:

1. >20 weeks gestation by best obstetrical estimate
2. Post partum and not anticipating another pregnancy within 18 months
3. Preconception and not anticipating another pregnancy within 18 months
4. Not cognitively aware enough to participate in the study
5. Not willing to undergo at least two periodontal exams
6. <18 years of age
7. Not willing to chew 1 piece of xylitol gum for 10 minutes after the morning and evening meal (intervention sites)
8. Anticipating a move outside of the region within 18 months

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10069 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Aagaard, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment through outpatient prenatal clinics
Pre-assignment Details: All patients who were eligible and consented for the study were enrolled and designated into either a control or intervention group based on this cluster-randomized design and the site of enrollment where the participant initially presented.
Units Other Than Participants: 8
Period: Overall Study
Arm/Group | Control | Xylitol
Started (Enrolled and consented to the PPaX trial) | 5520; 4 8 | 4549; 4 8
Completed (Analyzed for primary outcomes) | 5321; 4 8 | 4349; 4 8
Not Completed | 199; 0 8 | 200; 0 8
Not completed — Lost to Follow-up | 137 | 106
Not completed — Pregnancy Interrupted | 42 | 89
Not completed — Enrolled prepregnant without neonatal outcome data available | 20 | 5

BASELINE CHARACTERISTICS:
Population: Includes 10069 total individuals who were eligible and enrolled in the PPaX trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Xylitol | Total
Number analyzed (Participants) | 5520 | 4549 | 10069
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5520 | 4549 | 10069
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5520 | 4549 | 10069
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African, black | 5520 | 4549 | 10069
Region of Enrollment [Number; unit: participants]
  Malawi | 5520 | 4549 | 10069

OUTCOME MEASURES:

1. Primary Outcome: Rate of Preterm Birth
Description: This is a co-primary outcome: Measure rate of preterm birth <37 weeks gestation, as defined by best obstetrical estimate based upon last menstrual period correlated with fundal height at entry to prenatal care or ultrasound, when available; all sites have access to referral for ultrasound.
Time Frame: Conception to date of delivery, <37 weeks gestation
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control group (no xylitol gum exposure)
- Xylitol: Intervention group (twice daily xylitol gum use during pregnancy)
Arm/Group | Control | Xylitol
Number analyzed (Participants) | 5321 | 4349
Participants | 878 | 549
Statistical Analysis 1: Comparison: Control vs Xylitol; Test type: Superiority; p < 0.05, Mixed Models Analysis; We employed generalized linear mixed methods (GLMM) with binomial distribution to examine the association between study primary outcomes of baby's birth weight (<2500) and gestational age at delivery (<37 weeks including up to 36 and 6/7 weeks) and assignment to the study intervention group. To account for clustering of outcomes by cluster (sites), we used random slope/random intercept GLMM models with a cluster as a random effect (level 2) and treatment as a fixed effect (level 1), since random effect modeling is an individual-level analyses that accounts for within-cluster dependence by maximum likelihood estimation. A separate model was fit to each study outcome and corresponding relative risk with 95% confidence intervals (CI) estimated. Full information maximum likelihood estimation (FIML) allows for analyses to be performed with the full sample, under conditions of Missing Completely at Random (MCAR) and Missing at Random (MAR), and with missing data rates up to 50%

2. Primary Outcome: Number of Infants <2500 Grams
Description: This is a co-primary outcome: Measured weight at delivery to determine the rate of <2500 gram infants.
Time Frame: Date of delivery to 1 week postnatal
Population: There were 5260 of the 5520 subjects in the control group after removing 42 with an interrupted pregnancy, 20 prepregnant without information on neonatal outcomes, 137 lost to follow up, and 61 with only neonatal gestational age information.
  There were 4305 of 4349 consented for enrollment in the xylitol intervention group, after removing 89 with an interrupted pregnancy, 5 prepregnant without neonatal outcomes data, 106 lost to follow up and 45 with only neonatal gestational age data.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Xylitol
Number analyzed (Participants) | 5260 | 4305
Participants | 679 | 385
Statistical Analysis 1: Comparison: Control vs Xylitol; Co-primary outcomes; Test type: Superiority; p < 0.05, Mixed Models Analysis; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Infants With Adverse Neonatal Composite Morbidity and Mortality
Description: Additive or singular composite neonatal morbidity up to 28 days of age. Composite neonatal morbidity and mortality outcomes are defined as: neonatal death, miscarriage <28 weeks, stillbirth (fresh or macerated), neonatal sepsis, neonatal respiratory distress, neonatal seizures, feeding problems, fever, hypothermia, Apgar score <7 at 5 minutes after birth, referral to other hospital or neonatal intensive care unit (NICU)
Time Frame: Date of delivery to 28 days postnatal
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Xylitol
Number analyzed (Participants) | 5321 | 4349
Participants | 238 | 133
Statistical Analysis 1: Comparison: Control vs Xylitol; Test type: Superiority; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Number of Participants With Periodontal Disease
Description: We will measure the prevalence of periodontal disease among gravidae. We will use standardized World Health Organization (WHO) oral health forms and disease scoring.
Time Frame: During pregnancy, up to 2 dental visits performed during pregnancy (approximately 37-40 weeks if term) to evaluate dental outcomes
Population: There were 461 subjects in the control group who completed at least 2 dental visits. There were 490 subjects in the intervention, xylitol group who completed at least 2 dental visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Xylitol
Number analyzed (Participants) | 461 | 490
Participants | 117 | 102
Statistical Analysis 1: Comparison: Control vs Xylitol; Test type: Superiority; p < 0.05, Mixed Models Analysis; Specifically, the composite of periodontal disease was also created; this composite was positive if any of the following were detected: gingival bleeding, pockets of 4 mm or greater, or loss of attachment of 4 mm or greater. A scaled periodontal disease score was also created which was the sum of scores for gingival bleeding (+1 if bleeding was present, per tooth), gingival pockets (+1 for pockets of 4-5 mm and +2 for 6 mm or deeper, per tooth), and loss of attachment (+1 for 4-5 mm loss, +2 for 6-8 mm, +3 for 9-11 mm, and +4 for 12 mm or more, per tooth with values recorded for index teeth) divided by the number of teeth present

5. Secondary Outcome: Number of Participants With Dental Caries
Description: We will measure the prevalence of dental caries among gravidae. We will use standardized World Health Organization (WHO) oral health forms and disease scoring.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Xylitol
Number analyzed (Participants) | 461 | 490
Participants | 123 | 135
Statistical Analysis 1: Comparison: Control vs Xylitol; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 4 years; Data was collected from study enrollment in 2015 through 2019 during which study participants were enrolled and completed the study. An additional 2 year follow-up period occurred from 2019-2021 in which data was verified and cross-validated with local maternal delivery logbooks
Arm/Group | Control | Xylitol
All-Cause Mortality (participants affected / at risk) | 2/5520 | 0/4549
Serious Adverse Events (participants affected / at risk) | 2/5520 | 0/4549
Other Adverse Events (participants affected / at risk) | 0/5520 | 0/4549
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=5520) | Xylitol (N=4549)
Death (Pregnancy, puerperium and perinatal conditions) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02333227/Prot_SAP_ICF_000.pdf